CLINICAL TRIAL: NCT01385826
Title: Evaluation of the Efficacy of Adalimumab for the Treatment of Uveitis in Juvenile Idiopathic Arthritis: Randomized Double-blind Placebo-controlled Trial
Brief Title: Effect of Adalimumab for the Treatment of Uveitis in Juvenile Idiopathic Arthritis
Acronym: ADJUVITE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Abbott (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P081210
Record Dates: First submitted 2011-05-24; First posted 2011-06-30 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Uveitis; Juvenile Arthritis
Keywords: Uveitis; Juvenile arthritis; Anti-tumor necrosis factor alpha monoclonal antibody; treatment
MeSH Terms: conditions — Uveitis; Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- adalimumab (Experimental): Anti-tumor necrosis factor alpha monoclonal antibody
  Interventions: Drug: Anti-tumor necrosis factor alpha monoclonal antibody
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Anti-tumor necrosis factor alpha monoclonal antibody — The dose of adalimumab will be 40 mg for children age 13 and over and for children younger than 13 adalimumab 24 mg per m2 BSA (up to a maximum total body dose of 40 mg).
  Arms: adalimumab
Drug: placebo — Patients will receive 4 injections of placebo on D0, D14, D28, and D42 with assessment of the primary endpoint at M2
  Arms: placebo

SUMMARY:
The investigators propose to study the efficacy of adalimumab versus placebo (double-blind randomization on inclusion into 2 equal groups) on reduction of ocular inflammation quantified by laser flare photometry after two months of treatment in patients with active uveitis despite well conducted treatment with steroid eye drops and MTX. The primary objective is to demonstrate a higher response rate at 2 months in the adalimumab arm versus the placebo arm. Will be considered as responding patients those in whom the evaluated eye, 2 months after inclusion, presents at least 30% reduction of inflammation on laser flare photometry and improvement or a stable appearance on slit lamp examination. After the second month, all patients wishing to continue the trial and presenting a satisfactory clinical state will be treated with adalimumab for a total of one year after inclusion to descriptively evaluate the efficacy and safety of treatment over 10 to 12 months.

DETAILED DESCRIPTION:
20% of patients with juvenile idiopathic arthritis (JIA) develop usually bilateral, chronic anterior uveitis, dependent on steroid eye drops and sometimes systemic steroid therapy, with a risk of complications such as cataract, band keratopathy and glaucoma, usually responsible for loss of vision. No maintenance treatment has been demonstrated to be effective. Methotrexate (MTX), the maintenance treatment most commonly used in JIA, could have a beneficial effect, but this effect is not sufficient to stop progression of uveitis in most patients. Our preliminary experience and that of other teams based on small series of patients is in favour of the efficacy of anti-Tumour Necrosis Factor alpha (TNFalpha) monoclonal antibodies (Ab) in JIA-associated uveitis. An international multicentre randomized trial of a humanized monoclonal antibody, adalimumab, in JIA has demonstrated its efficacy on joint lesions and its good safety as monotherapy or in combination with methotrexate. However, children with active uveitis were excluded from this trial.

The investigators propose a French multicentre, randomized, double-blind, placebo-controlled trial to evaluate the efficacy of adalimumab in JIA-associated uveitis in patients over the age of 4 years. These patients must have active uveitis (Laser flare-cell meter score of at least 30 photons/ms) despite topical steroid therapy, with intolerance or failure to at least 3 months of MTX therapy. The dose of adalimumab will be 40 mg eow for children age 13 and over and for children younger than 13 adalimumab 24 mg per m2 BSA (up to a maximum total body dose of 40 mg). The activity of uveitis will be evaluated by laser flare photometry, a recently validated technique for follow-up of the efficacy of treatments of anterior uveitis. Seven hospital ophthalmology departments in France are equipped with laser flare photometry and have a sufficient experience to participate in this trial (Paris-Pitie-Salpetriere, Paris-Cochin, Nantes, Lille, Grenoble, Bordeaux and Lyon). Several teams of paediatric rheumatologists and hospital rheumatologists working with these ophthalmology departments will also be able to include patients. The primary endpoint is an at least 30% reduction of ocular inflammation after 2 months of treatment, quantified by laser flare photometry, considering the more severely affected eye in the case of bilateral uveitis. Based on the hypothesis of a response rate of at least 50% with adalimumab versus a maximum of 10% with placebo, comparison of two groups of 19 patients would be sufficient to conclude on a significant difference for a two-sided alpha risk of p=0.05 and a power of 80%. The investigators therefore plan to include 40 patients with randomization to two equal groups, one receiving 4 subcutaneous injections of adalimumab and the other receiving 4 injections of placebo on D0, D14, D28, and D42 with assessment of the primary endpoint at M2. The planned duration of inclusion is 2 years with a total duration of the trial of 3 years. From visit M2 onwards, all patients will be treated by adalimumab injections every 2 weeks and will be followed for 1 year of treatment. Clinical, laboratory and ophthalmological evaluation including laser flare photometry and conventional slit lamp examination will be performed at each visit (pre-inclusion, D0, D14, M1, M2, M3, M4, M5, M6, M9 and M12). Deterioration of ocular inflammation during the first 2 months will justify decoding for the patient concerned who will be considered to be a treatment failure.

A study will be conducted in parallel: gene expression profile studies on whole blood by a team experienced in the study of JIA and other inflammatory diseases (Dr Pascual, Dallas, USA).

ELIGIBILITY:
Inclusion Criteria:

1. Active uveitis associated with juvenile idiopathic arthritis, with the exclusion of systemic JIA, juvenile-onset rheumatoid arthritis, and enthesitis-related JIA
2. Uveitis resistant to well conducted topical steroid therapy comprising either dexamethasone or rimexolone at a dose adapted to the patient's situation as validated by one of the investigating ophthalmologists.
3. Failure of systemic treatment with methotrexate at a dose of 0.3 to 0.6 mg.kg (without exceeding 25 mg) once a week for at least 3 months (except in the case of methotrexate intolerance).
4. Patient who can be evaluated by laser flare photometry.
5. Patient at least 4 years old on initiation of trial medication and weighing a minimum of 15 kg
6. Signed informed consent both parents and/or patient's agreement
7. Patient has a social security or similar

Exclusion Criteria:

1. Systemic JIA, juvenile-onset rheumatoid arthritis, enthesitis-related JIA (with a risk of red eye uveitis).
2. History of treatment with anti-TNF alpha monoclonal antibody (either adalimumab or infliximab).
3. Any contraindication to administration of immunosuppressive therapy (immune deficit, opportunistic infection, other severe chronic disease)

   * History of cancer or lymphoproliferative disease other than successfully and completely resected squamous cell or basal cell skin cancer,
   * Any uncontrolled disease: unstable diabetes with documented history of recurrent infections, unstable ischaemic heart disease, moderate to severe heart failure (NYHA stage III/IV), recent stroke and any other disease or condition inducing, in the investigator's opinion, a risk for the patient related to his/her participation in the trial,
   * Positive hepatitis B or C serology indicating active infection,
   * History of positive HIV serology,
   * Persistent infection or severe infections requiring hospitalisation or IV antibiotic therapy during the 30 days prior to inclusion in the trial or oral antibiotic therapy during the 14 days prior to inclusion in the trial,
   * History of clinically significant alcohol or other substance abuse during the previous year,
   * Previous diagnosis or signs of demyelinating disease of the central nervous system,
   * History of active tuberculosis, histoplasmosis or listeriosis,
   * Signs of latent tuberculosis (based on a history of nontreated contamination, or an opacity greater than 1 cm on chest x-ray, or a positive intradermal reaction to 5 IU of tuberculin ≥ 5 mm).
   * Negative urine pregnancy test in girls with childbearing potential
4. Chronic rupture of the blood-aqueous barrier with marked flare on the initial examination but not modified by one month of anti-inflammatory therapy.
5. Impossibility to monitor flare:

   * Children < 4 years
   * False flare due to the presence of giant cells on the surface of an artificial lens or in an aphakic child.
6. Children presenting complications such as refractory glaucoma or cataract rapidly requiring surgery.
7. Phthisis bulbi with hypotonia and atrophy of the ciliary body.
8. Any other situation raising problems for maintenance of stable doses of steroids and immunosuppressive drugs during the period between 4 weeks before D0 and the M2 evaluation. Authorized immunosuppressive therapies that must be maintained at stable dose are steroid eye drops, systemic steroid therapy and once weekly oral or subcutaneous MTX at a dose of 0.3 to 0.6 mg (without exceeding 25 mg).
9. Any ophthalmologic contraindication
10. If female and childbearing potential should have an appropriate contraceptive method during all study period and 5 months after last adalimumab dose. Abstinence with no oral contraception can be considered.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-06-29 (Actual); Primary Completion 2014-11-04 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
To demonstrate that a higher proportion of subjects will have an improvement of uveitis on adalimumab versus placebo after 2 months relative to baseline | Final visit could occur at any point up to 78 weeks
  The primary objective is to demonstrate the efficacy of 2 months of treatment with adalimumab versus placebo on reduction of ocular inflammation in JIA-associated uveitis.
  By defining response to treatment as a reduction of at least 30% of ocular inflammation quantified by laser flare photometry in the initially more severely inflamed eye without deterioration of cell count or flare protein on slit lamp examination, we formulate the hypothesis that at least 50% of patients treated with adalimumab for 2 months will respond to treatment versus a maximum 10% of patients on placebo.

SECONDARY OUTCOMES:
Evaluation of adverse events | 12 months
  To evaluate the safety of treatment at 2 months then at 12 months
Proportion of subjects at each study time point with an improvement of uveitis | 2 months
  To evaluate the response of the treatment on ocular inflammation quantified by slit lamp examination and laser flare photometry at each visit comparatively between the adalimumab arm and the placebo arm during the double-blind period (until M2, as a complement to the laser flare photometry evaluation performed for the primary objective) and then descriptively on adalimumab. Analyses will be performed on the eye evaluated for the primary objective and for the fellow eye in patients with bilateral uveitis.
Eyes with active uveitis | 2 months
  To compare the proportion of eyes with active uveitis on inclusion improved after 2 months between the adalimumab arm and the placebo arm
The efficacy of treatment on juvenile idiopathic arthritis | 2 months
  To evaluate the efficacy of treatment on JIA, particularly the joint lesions at each visit, comparatively between the adalimumab arm and the placebo arm until M2 then descriptively on adalimumab
Decrease topical or systemic steroid therapy | 12 months
  To evaluate the possibility to decrease topical steroid therapy and when applicable systemic steroid therapy between M2 and M12
Transcriptome modifications on whole blood | 12 months
  To evaluate possible transcriptome modifications on whole blood in the context of a collaboration with a team experienced in analysis of cytokine signatures associated with JIA and other inflammatory diseases in children (team directed by V. Pascual in Dallas).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Quartier dit Maire, MD, PhD, Principal Investigator — hospital Necker Enfants Malades
Locations (1):
- Hospital of necker Enfants malades, Paris, France

REFERENCES:
- [Background] Quartier P, Baptiste A, Despert V, Allain-Launay E, Kone-Paut I, Belot A, Kodjikian L, Monnet D, Weber M, Elie C, Bodaghi B; ADJUVITE Study Group. ADJUVITE: a double-blind, randomised, placebo-controlled trial of adalimumab in early onset, chronic, juvenile idiopathic arthritis-associated anterior uveitis. Ann Rheum Dis. 2018 Jul;77(7):1003-1011. doi: 10.1136/annrheumdis-2017-212089. Epub 2017 Dec 23. PMID 29275333
- [Background] Simonini G, Taddio A, Cattalini M, Caputo R, De Libero C, Naviglio S, Bresci C, Lorusso M, Lepore L, Cimaz R. Prevention of flare recurrences in childhood-refractory chronic uveitis: an open-label comparative study of adalimumab versus infliximab. Arthritis Care Res (Hoboken). 2011 Apr;63(4):612-8. doi: 10.1002/acr.20404. PMID 21452272
- [Background] Callejas-Rubio JL, Sanchez-Cano D, Serrano JL, Ortego-Centeno N. Adalimumab therapy for refractory uveitis: a pilot study. J Ocul Pharmacol Ther. 2008 Dec;24(6):613-4; author reply 614. doi: 10.1089/jop.2008.0073. No abstract available. PMID 19049264
- [Background] Tynjala P, Kotaniemi K, Lindahl P, Latva K, Aalto K, Honkanen V, Lahdenne P. Adalimumab in juvenile idiopathic arthritis-associated chronic anterior uveitis. Rheumatology (Oxford). 2008 Mar;47(3):339-44. doi: 10.1093/rheumatology/kem356. Epub 2008 Jan 31. PMID 18238789
- [Background] Biester S, Deuter C, Michels H, Haefner R, Kuemmerle-Deschner J, Doycheva D, Zierhut M. Adalimumab in the therapy of uveitis in childhood. Br J Ophthalmol. 2007 Mar;91(3):319-24. doi: 10.1136/bjo.2006.103721. Epub 2006 Oct 11. PMID 17035274
- [Background] Vazquez-Cobian LB, Flynn T, Lehman TJ. Adalimumab therapy for childhood uveitis. J Pediatr. 2006 Oct;149(4):572-5. doi: 10.1016/j.jpeds.2006.04.058. PMID 17011337